CLINICAL TRIAL: NCT06533241
Title: Trends of Renal Biopsy in Pediatric Patients at Tanta University Hospital
Brief Title: Trends of Renal Biopsy in Pediatric Patients at Tanta University Hospital for 10 Years From 2012 to 2022.
Status: Active, not recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, Principal Investigator, Clinical Lecturer of Pediatric Nephrology, Tanta University
Other Study IDs: 36264PR419/11/23
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Renal Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients less than 18 years' old who underwent renal biopsy: pediatric patients less than 18 years' old who underwent renal biopsy at Tanta University Hospital from 2012 to 2022.
  Interventions: Procedure: renal biopsy

INTERVENTIONS:
Procedure: renal biopsy — percutaneous renal biopsy procedure

SUMMARY:
This study will be conducted on pediatric patients less than 18 years' old who underwent renal biopsy at Tanta University Hospital from 2012 to 2022.

DETAILED DESCRIPTION:
This study will be conducted on pediatric patients less than 18 years' old who underwent renal biopsy at Tanta University Hospital from 2012 to 2022.

The data will be collected from records:

1. History taking including age and sex.
2. Indications for renal biopsy.
3. Methods of renal biopsy
4. Complications of renal biopsy
5. Adequacy of samples
6. The results obtained by light microscopy
7. The results obtained by electron microscopy, immunofluorescence when indicated

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients less than 18 years' old who underwent renal biopsy.

Exclusion Criteria:

* no exclusions

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients less than 18 years' old who underwent renal biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
the indications of renal biopsy | 3 months
  investigate the indications of renal biopsy in pediatric patients at Tanta University Hospital for 10 years from 2012 to 2022

SECONDARY OUTCOMES:
light , electron microscope and immunofluorescence results of renal biopsy | 3 months
  investigate the results of renal biopsy in pediatric patients at Tanta University Hospital for 10 years from 2012 to 2022

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mabrouk Mohamed Elghoul, MD, Principal Investigator — Tanta University
Locations (1):
- Sara Mabrouk Mohamed Elghoul, Tanta, Tanta, Qism 1, Egypt

IPD SHARING:
Plan to Share IPD: Undecided